CLINICAL TRIAL: NCT06279533
Title: Safety and Pharmacokinetics Study of Multiple Ascending Doses and Food Effect of LV232 Capsules in Chinese Healthy Volunteers
Brief Title: Safety and Pharmacokinetics Study of Multiple Ascending Doses and Food Effect of LV232 Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vigonvita Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LV232-02
Record Dates: First submitted 2024-01-31; First posted 2024-02-28 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-02

CONDITIONS: Healthy Subjects
Keywords: LV232; Phase I; dose-escalation; Tolerability; Pharmacokinetic; food effect

STUDY DESIGN:
Intervention Model Description: PK characteristics of multiple ascending doses study is parallel design, and FE study is crossover design
Who Masked: Participant, Care Provider, Investigator
Masking Description: PK characteristics of multiple ascending doses study is double-blinded, placebo-controlled design, and FE study is open-label design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PK characteristics of multiple ascending doses study (Experimental): There are 24 subjects devided into 3 dose groups (15mg, 40mg and 60mg).8 subjects will be enrolled in each dose group and the ratio of investigational product to placebo is 3:1. LV232/Placebo is administered sequentially from low-dose to high-dose and each subject can only orally receive one dose level. Investigational product is orally administrated QD for day1, day3~day9. When 7th day visit after last dose (D15) is completed for previous dose group, investigator and sponsor will evaluate the safety and determine whether the next dose group can be started or adjusted.
  Interventions: Drug: LV232/Placebo
- FE study (Experimental): 24 healthy subjects divided into 2 group (20mg and 60mg) will be enrolled once all eligibility criteria are met after screening within 14 days prior to investigation product administration. Informed consent should be obtained before any protocol defined procedures can be started.Investigational product administration plan given below: 12 healthy subjects in each group will be randomized to 3 sub-groups, i.e., Group A, Group B, Group C, with 4 subjects in each sub-group. For group A, investigation product will be given after fasting for Period 1, after standard diet for Period 2, and after high-fat diet for Period 3; For group B, investigation product will be given after high-fat diet for Period 1, after fasting for Period 2, and after standard diet for Period 3; For group C, investigation product will be given after standard diet for Period 1, after high-fat diet for Period 2, and after fasting for Period 3. Wash-out period is 5 days.
  Interventions: Drug: LV232

INTERVENTIONS:
Drug: LV232/Placebo — Drug: LV232 15mg Group:
  6 subjects will receive LV232 15mg, orally; Other Names:Placebo 2 subjects will receive placebo, orally.
  Drug: LV232 40mg Group:
  6 subjects will receive LV232 40mg, orally; Other Names:Placebo 2 subjects will receive placebo, orally.
  Drug: LV232 60mg Group:
  6 subjects will receive LV232 60mg, orally; Other Names:Placebo 2 subjects will receive placebo, orally.
  Other Names: LV232 15mg; LV232 40mg; LV232 60mg
  Arms: PK characteristics of multiple ascending doses study
Drug: LV232 — Drug: LV232 20mg Group:
  12 subjects will receive LV232 20mg, orally
  Drug: LV232 60mg Group:
  12 subjects will receive LV232 60mg, orally
  Other Names: LV232 20mg; LV232 60mg
  Arms: FE study

SUMMARY:
This study is divided into two parts: the safety, tolerability, pharmacokinetic profiles of LV232 capsules after multiple ascending doses (hereinafter referred to as "PK characteristics of multiple ascending doses study ") and food effect study (hereinafter referred to as "FE study"). A total of 48 subjects are planned to be enrolled. The two parts of the study can be carried out simultaneously, and there is no order requirement.

DETAILED DESCRIPTION:
PK characteristics of multiple ascending doses study is used randomized, double-blinded, placebo-controlled, single-center design. LV232/Placebo is administered sequentially from low-dose to high-dose and each subject can only orally receive one dose level. There are 3 dose groups (15mg, 40mg and 60mg), 8 subjects will be enrolled in each dose group and the ratio of investigational product to placebo is 3:1. Investigational product is orally administrated QD for day1, day3~day9. When 7th day visit after last dose (D15) is completed for previous dose group, investigator and sponsor will evaluate the safety and determine whether the next dose group can be started or adjusted.

FE study is a single-center, randomized, open-label, three-period crossover design. 24 healthy subjects divided into 2 groups (20mg、60mg) will be enrolled once all eligibility criteria are met after screening within 14 days prior to investigation product administration. Informed consent should be obtained before any protocol defined procedures can be started.Investigational product administration plan given below: 12 healthy subjects in each group will be randomized to 3 sub-groups, i.e., Group A, Group B, Group C, with 4 subjects in each sub-group. For group A, investigation product will be given after fasting for Period 1, after standard diet for Period 2, and after high-fat diet for Period 3; For group B, investigation product will be given after high-fat diet for Period 1, after fasting for Period 2, and after standard diet for Period 3; For group C, investigation product will be given after standard diet for Period 1, after high-fat diet for Period 2, and after fasting for Period 3. The wash-out period is 5 days.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 45 years old, males or females;
2. Body weight no less than 50.0 kg for male, no less than 45.0 kg for female,Body Mass Index of 19.0 to 26.0kg/m2;
3. Physical examination, vital signs examination, laboratory examination, electrocardiogram examination and B-ultrasound examination results were normal or abnormal without clinical significant;
4. Subjects who are willing to take effective contraceptive during the study and within 3 months after the study completed;
5. Subjects who are able to understand and follow study plans and instructions; Subjects who have voluntarily decided to participate in this study, and signed the informed consent form.

Exclusion Criteria:

1. Subjects with hypersensitivity to LV232 or any of the excipients;
2. Subjects with allergic diseases or allergic constitution;
3. Subjects with skin diseases or a history of skin allergies;
4. Subjects with central nervous system, cardiovascular system, gastrointestinal, respiratory system, urinary, Hematologic System, metabolic disorders that require medical intervention or other diseases (such as psychiatric history) that are not suitable for clinical trials;
5. Blood donation or blood loss ≥ 400 mL within 3 months , or have a history of blood product use history
6. Subjects who have participated in clinical trials of other drugs within 3 months before screening;
7. Subjects who have taken any prescription drugs, over-the-counter drugs, Chinese herbal medicines, or health products orally within 2 weeks before screening;
8. Drug or alcohol addicts within 1 year prior to screening, who drink at least twice a day or more than 14 units per week, or who are addicted to alcohol (1 unit ≈200 mL beer with 5% alcohol content, 25 mL spirits with 40% alcohol content or 85 mL wine with 12% alcohol content);
9. Subjects who smoked more than 10 cigarettes or equivalent amounts of tobacco a day within one year before screening;
10. Subjects who can't quit smoking and drinking during the experiment;
11. Subjects who are positive for hepatitis B virus surface antigen, hepatitis C virus antibody, Treponema pallidum antibody (TPPA) or human immunodeficiency virus antibody (Anti-HIV);
12. Abnormal and clinically significant chest radiographs (anteroposterior);
13. B ultrasound examination showed moderate to severe fatty liver;
14. Pregnant or lactating woman or male subjects whose spouse has a child care plan within 3 months;
15. The investigator believes that there are other factors that are not suitable for participating in this trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Tmax | Calculated using concentration data collected from predose to 72 hours postdose
  Maximum observed plasma concentration
Cmax | Calculated using concentration data collected from predose to 72 hours postdose
  Maximum observed plasma concentration
T1/2 | Calculated using concentration data collected from predose to 72 hours postdose
  Terminal half life
AUC0-t | Calculated using concentration data collected from predose to 72 hours postdose
  Area under the serum concentration time profile from time zero to the time of the last quantifiable concentration
AUC0-24h | Calculated using concentration data collected from predose to 24 hours postdose
  Area under the serum concentration time profile from time zero to the time of 24h
AUC0-∞ | Calculated using concentration data collected from predose to 72 hours postdose
  Area under the plasma concentration-time curve from time 0 extrapolated to infinity

SECONDARY OUTCOMES:
Number of participants with treatment emergent treatment-related adverse event(s) | Dosing through follow-up call (7 days after last dose of investigational product)
  Frequency, severity and causal relationship of treatment emergent adverse events
Laboratory test | Dosing through follow-up call (7 days after last dose of investigational product)
  Number of participants with laboratory test findings of potential clinical importance
Vital signs | Dosing through follow-up call (7 days after last dose of investigational product)
  Number of participants with vital signs findings of potential clinical importance
Number of participants with ECG findings of potential clinical importance | Dosing through follow-up call (7 days after last dose of investigational product)
  Number of subjects with change from baseline in electrocardiogram (ECG) parameters

CONTACTS AND LOCATIONS:
Overall Officials: Chen Yu, Principal Investigator — Shanghai Xuhui Central Hospital
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, China